CLINICAL TRIAL: NCT02361398
Title: Individualized Positive End Expiratory Pressure(PEEP) Setting by EIT in Patients With Acute Respiratory Distress Syndrome(ARDS)
Brief Title: Individualized PEEP Setting by EIT in Patients With ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-ARDS-EIT
Record Dates: First submitted 2015-01-13; First posted 2015-02-11 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: the PEEP Setting of ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT group (Experimental): the Individualized PEEP titration by EIT was administered to the patients in the EIT group.
  Interventions: Other: the EIT guide the individualized PEEP Setting
- control group (No Intervention): If patients are assigned to the control group, the Individualized PEEP Setting was by PEEP-FiO2 table based on ARDS-net protocol.

INTERVENTIONS:
Other: the EIT guide the individualized PEEP Setting — the EIT guide the individualized PEEP Setting in the EIT group
  Arms: EIT group

SUMMARY:
The investigators conducted a pilot study to compare the effect of Positive End Expiratory Pressure(PEEP) setting guide by lung electrical impedance tomography(EIT) and ARDS-net PEEP-FiO2 table on survival in subjects with mild/severe Acute Respiratory Distress Syndrome(ARDS).

ELIGIBILITY:
Inclusion:

1. acute respiratory distress syndrome with ratio of partial pressure of arterial oxygen over fraction of inspired oxygen (PaO2:FiO2)<300 and PEEP >5cmH2O
2. Body mass index < =40
3. Written inform consent

Exclusion:

1. pregnant，intracranial hypertension
2. left ventricular dysfunction (EF<25% )
3. Patients with end-stage conditions(death expected within 90 days)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
survival | 28-day
  Non-survive and survive
Arterial oxygenation | 72h
  PaO2(mmHg) measured by blood gas analysis

SECONDARY OUTCOMES:
length of ICU stay and mechanical ventilated day | 28days
  Days of ICU stay and received mechanical ventilation(day)
pneumothorax requiring chest tube during first 7 days; barotrauma during first 7 days; | 7days
  new-onset of pneumothorax and barotrauma

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Director — Department of Critical Care Medicine, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences,, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] He H, Chi Y, Yang Y, Yuan S, Long Y, Zhao P, Frerichs I, Fu F, Moller K, Zhao Z. Early individualized positive end-expiratory pressure guided by electrical impedance tomography in acute respiratory distress syndrome: a randomized controlled clinical trial. Crit Care. 2021 Jun 30;25(1):230. doi: 10.1186/s13054-021-03645-y. PMID 34193224